CLINICAL TRIAL: NCT02531061
Title: Impact of the Persistence of Inflammation at Doppler Ultrasound Level on the Structural Evolution of Erosion in Rheumatoid Arthritis Treated With Biotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1208092; 2012-A01583-40 (Other: ANSM)
Record Dates: First submitted 2015-08-20; First posted 2015-08-21 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; bDMARDs; biotherapy; remission; erosion
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- active erosion (Experimental): HR-pQCT for measure bone parameters in "active erosion" group. The "active erosion" group will be defined by grades 2 and 3, ie by the presence of Doppler signals confluence in less than 50% of the synovial surface (grade 2) and in over 50% of the surface synovial for grade 3
  Interventions: Device: HR-pQCT
- inactive erosion (Experimental): HR-pQCT for measure bone parameters in "active erosion" group. The "inactive erosion" group will be defined by grades 0 and 1, ie the absence of Doppler signal for grade 0 and the presence of some non confluence Doppler signals for the grade 1
  Interventions: Device: HR-pQCT

INTERVENTIONS:
Device: HR-pQCT — The Xtrem CT scanco device is a HR-pQCT. It was initially used to measure bone density and quantify the bone architecture to 3D at the extremities of the human body.
  For the study, the device will be used to measure changes in erosion at the 2nd or 3rd metacarpal head. Only the patient's hand will be in contact with the medical device, the acquisition time will be 3 minutes.
  Other Names: Xtrem CT scanco

SUMMARY:
Since biological disease-modifying anti-rheumatic drugs (bDMARDs) are available in rheumatoid arthritis (RA) strategy an emerging question is the definition of remission in RA. Today some criteria were already proposed and the last one was proposed in 2011.

All these criteria integrated only clinical criteria without imaging assessment. In this context, ultrasound joint is daily performed without definition of remission. A discrepancy exists between clinical remission and persistence of active disease with ultrasound joint presence of a Doppler effect indicating inflammation and the risk of progression of joint damage. A definition of remission in RA could include erosions regression in subchondral bone (at best measured by high resolution peripheral quantitative computed tomography (HR-pQCT)).

The main hypothesis is that the reduction of erosion size assessed by HR-pQCT will be observed only in the absence of local inflammation measured by Doppler ultrasound in the erosion.

Tumor Necrosis Factor (TNF) blockers have strongly improved RA therapy outcome in terms of clinical improvement and structural damage (progression of radiographic lesions). Recent data showed that there could be joint bone rebuilt in case of inflammation suppression. HR-pQCT is a new technique emerging for bone erosions assessment in RA. Erosions size and volume could be reduced with anti-TNF, but with a large interindividual variability. There was no correlation between the activity of clinical or ultrasound synovium and evolution of erosion HR-pQCT.

ELIGIBILITY:
Inclusion Criteria:

* Initial medical examination performed,
* RA diagnosis according to the criteria of the ACR / EULAR 2010
* Low or moderate disease activity with a DAS28 ≤ 4 since at least for 6 months
* Patients with bDMARDs (Remicade®, Enbrel®, Humira®, Cimzia®, Simponi®, Ro-Actemra®, ou Orencia®) since at least 6 months and no change planned by the investigator,
* Patient with at least one erosion on the head of the 2nd or 3rd metacarpal right or left,
* Stable corticosteroids dose since at least 3 months less than or equal to 10 mg of prednisone equivalent,
* Medical care and monitoring in the rheumatology department of the CHU of Saint-Etienne or the Edouard Herriot Hospital in Lyon,
* written consent of patient

Exclusion Criteria:

* Other diagnosis than RA,
* Intravenous or intra-articular injection at the 2nd or 3rd metacarpophalangeal left or right during the 3 months prior to inclusion,
* Surgery provided at the 2nd or 3rd metacarpophalangeal right or left within a year of inclusion,
* Concomitant treatment with zoledronic acid (Aclasta) or denosumab (Prolia®)
* Refusal of blood collection,
* Pregnancy or breastfeeding women,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-05-05 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Change in depth of the erosion | baseline from 1 year
  compare the change in the depth of the erosion of the second or third metacarpal head right or left at 12 months between patients with "active erosion" and those with "inactive erosion" in RA patients with low disease activity treated with bDMARD since at least 6 months (Remicade®, Enbrel®, Humira®, Cimzia®, Simponi®, Ro-Actemra®, or Orencia®).

SECONDARY OUTCOMES:
Change in volume of erosion | baseline from 1 year
  compare the change in volume of erosion of the second or third metacarpal head right or left at 12 months between patients with "active erosion" and those with "inactive erosion" in RA patients with low disease activity treated with bDMARD since at least 6 months (Remicade®, Enbrel®, Humira®, Cimzia®, Simponi®, Ro-Actemra®, or Orencia®).
Change in width of erosion | baseline from 1 year
  compare the change in width of erosion of the second or third metacarpal head right or left at 12 months between patients with "active erosion" and those with "inactive erosion" in RA patients with low disease activity treated with bDMARD since at least 6 months (Remicade®, Enbrel®, Humira®, Cimzia®, Simponi®, Ro-Actemra®, or Orencia®).
Change in density parameter of bone microarchitecture | baseline from 1 year
  compare the change in density parameter of bone microarchitecture of erosion of the second or third metacarpal head right or left at 12 months between patients with "active erosion" and those with "inactive erosion" in RA patients with low disease activity treated with bDMARD since at least 6 months (Remicade®, Enbrel®, Humira®, Cimzia®, Simponi®, Ro-Actemra®, or Orencia®). Density parameter of bone microarchitecture is a composite outcome : Total mineral volumetric density (mg/ccm HA), Trabéculaire mineral volumetric density (mg/ccm HA), Cortical mineral volumetric density (mg/ccm HA), Trabecular Number (1/mm), Trabecular thickness (mm), Trabecular Separation (mm), Mean distance between trabeculae (mm), Presence of new erosions and volume

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Marotte, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (2):
- France (2):
  - HCL - Hôpital EdouarD Herriot, Lyon
  - CHU Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No